CLINICAL TRIAL: NCT01128153
Title: A 24-week, Multicentre, Randomised, Double-Blind, Placebo-Controlled Phase IIIb Study to Evaluate Efficacy and Safety of Saxagliptin in Combination With Metformin and Sulfonylurea in Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control With Combination of Metformin and Sulfonylurea
Brief Title: Saxagliptin Triple Oral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680L00006; CV181-117
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Inadequate Glycaemic Control; Saxagliptin; Metformin; Sulfonylurea; Triple Oral Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin 5 mg once daily (Experimental)
  Interventions: Drug: Saxagliptin
- Placebo once daily (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — 5 mg tablet once daily for 24 weeks to be taken orally
  Other Names: Onglyza
  Arms: Saxagliptin 5 mg once daily
Drug: Placebo — tablet once daily for 24 weeks to be taken orally
  Arms: Placebo once daily

SUMMARY:
The purpose of this study is to determine whether the addition of saxagliptin to a patient's combination treatment of metformin and sulfonylurea for a 24 week period will provide better control of the patient's type 2 diabetes and will be well tolerated.

DETAILED DESCRIPTION:
A 24-week, Multicentre, Randomised, Double-Blind, Placebo-Controlled Phase IIIb Study to Evaluate Efficacy and Safety of Saxagliptin in Combination with Metformin and Sulfonylurea in Subjects with Type 2 Diabetes who have Inadequate Glycaemic Control with Combination of Metformin and Sulfonylurea

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Males or females with type 2 diabetes with inadequate glycaemic control (HbA1c > or = 7% and < or = 10%) despite being on combination of metformin and sulfonylurea for at least 8 weeks prior to Visit 1
* BMI < or = 40 kg/m2

Exclusion Criteria:

* Symptoms of poorly controlled diabetes including but not limited to marked polyuria and marked polydipsia with > 10% weight loss in 3 months prior to entry, or other signs and symptoms
* History of diabetic ketoacidosis or hyperosmolar non-ketotic coma
* Current or prior use within 3 months of Visit 1 of insulin, DDP4 inhibitor, GLP-1 analogues, and/or other oral anti-diabetic agents (other than metformin or sulfonylurea)
* Treatment with CYP3A4 inducers and/or potent CYP3A4/5 inhibitor
* Estimated CrCl < 60 ml/min at Visit 2
* CHF (NYHA class III or IV) and/or LVEF <40%
* Active liver disease and/or significant abnormal liver function defined as AST and/or ALT > 3 x ULN and/or bilirubin > 2.0 mg/dL at Visit 2.
* Creatine kinase > or = 10 x ULN at Visit 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayanti Visvanthan, MD, Study Chair — AstraZeneca; Simon Fisher, MD, Study Chair — AstraZeneca; Vinod Mattoo, MD, Study Chair — Bristol-Myers Squibb; Robert Moses, MBBS, Principal Investigator — Sydney Diabetes Centre
Locations (33):
- Australia (7):
  - Research Site, Broadmeadow, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Daw Park, South Australia
  - Research Site, Elizabeth Vale, South Australia
  - Research Site, Melbourne, Victoria
  - Research Site, Camperdown
  - Research Site, Herston
- Canada (4):
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Sydney Mines, Nova Scotia
  - Research Site, Thornhill, Ontario
  - Research Site, Kensington, Prince Edward Island
- India (5):
  - Research Site, Karnāl, Haryana
  - Research Site, Bangalore, Karnataka
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Pune, Maharashtra
  - Research Site, Coimbatore, Tamil Nadu
- South Korea (4):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Goyang, Kyounggi-do
  - Research Site, Daegu
  - Research Site, Seoul
- Research Site, Bangkok, Thailand
- United Kingdom (12):
  - Research Site, Reading, Berks
  - Research Site, Ely, Cambridgeshire
  - Research Site, Whitstable, Kent
  - Research Site, Westbury, Wiltshire
  - Research Site, Ashford
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Peterborough
  - Research Site, Wellingborough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the study from 35 centres in 6 countries (Australia, United Kingdom, Canada, Korea, India and Thailand). Participants were recruited between June 2010 and December 2010.
Pre-assignment Details: Participants were screened over 2 week period. 383 participants enrolled; 126 excluded (11 declined, 114 did not meet eligibility criteria, 1 lost to follow up).
Groups:
- SAXAGLIPTIN: Saxagliptin 5 mg tablet once daily for 24 weeks to be taken orally
- PLACEBO: Placebo tablet once daily for 24 weeks to be taken orally
Period: Overall Study
Arm/Group | SAXAGLIPTIN | PLACEBO
Started | 129 (Randomised) | 128 (Randomised)
Full Analysis Set | 127 (Received at least 1 dose of investigational product during 24 week blinded period) | 128 (Received at least 1 dose of investigational product during 24 week blinded period)
Completed | 113 (Completed 24 weeks) | 113 (Completed 24 weeks)
Not Completed | 16 | 15
Not completed — Adverse Event | 1 | 3
Not completed — Condition under investigation worsened | 8 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Incorrect enrolment to study | 2 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Developed discontinuation criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAXAGLIPTIN | PLACEBO | Total
Number analyzed (Participants) | 129 | 128 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.55) | 56.8 (11.49) | 57.0 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 80 | 74 | 154
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 59 | 57 | 116
  Asian | 70 | 71 | 141
Region of Enrollment [Number; unit: Participants]
  Australia | 25 | 25 | 50
  Canada | 10 | 10 | 20
  India | 35 | 34 | 69
  Korea, Republic of | 25 | 24 | 49
  Thailand | 8 | 10 | 18
  United Kingdom | 26 | 25 | 51
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.4 (5.26) | 29.1 (4.93) | 29.2 (5.09)
HbA1c [Mean (Standard Deviation); unit: %] | 8.38 (0.856) | 8.19 (0.832) | 8.28 (0.848)
2-hour Postprandial Glucose [Mean (Standard Deviation); unit: mg/dL] | 269.18 (76.814) | 265.6 (69.713) | 267.39 (73.220)
2-hour Postprandial glucose [Mean (Standard Deviation); unit: mmol/L] | 14.94 (4.263) | 14.74 (3.869) | 14.84 (4.064)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 162.24 (47.322) | 155.45 (38.37) | 158.84 (43.125)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.00 (2.626) | 8.63 (2.130) | 8.82 (2.393)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24, Last Observation Carried Forward (LOCF)
Description: Adjusted Mean Change in HbA1c from baseline to Week 24 using analysis of covariance model
Time Frame: From Baseline to Week 24 weeks
Population: Full Analysis Set which included all participants randomised to the study who received at least 1 dose of investigational product and who had a non-missing baseline value and at least 1 post-baseline measure. The full analysis set follows intention-to-treat principle.
Measure: Mean (95% Confidence Interval); unit: percent
Groups:
- Arm 1 - SAXAGLIPTIN: Saxagliptin 5 mg tablet once daily for 24 weeks to be taken orally
- Arm 2 - PLACEBO: Placebo tablet once daily for 24 weeks to be taken orally
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 127 | 127
percent | -0.74 [-0.89 to -0.60] | -0.08 [-0.23 to 0.07]
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-0.86 to -0.47], Standard Error of Mean 0.099 — Adjusted mean treatment difference from the ANCOVA model (Saxagliptin - Placebo)

2. Secondary Outcome: Change in 2-hour Postprandial Glucose (PPG) From Baseline to Week 24, Last Observation Carried Forward (LOCF) Measured as [mg/dL]
Description: Adjusted Mean Change in 2-hour PPG from baseline to Week 24 using analysis of covariance model
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 115 | 113
mg/dL | -11.66 [-23.38 to 0.07] | 5.08 [-6.45 to 16.60]
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p = 0.0301, ANCOVA; Mean Difference (Final Values) = -16.74, 95% CI 2-sided [-31.85 to -1.62], Standard Error of Mean 7.667 — Adjusted mean treatment difference from the ANCOVA model (Saxagliptin - Placebo)

3. Secondary Outcome: Change in 2-hour Postprandial Glucose (PPG) From Baseline to Week 24, Last Observation Carried Forward (LOCF) Measured as [mmol/L]
Description: Adjusted Mean Change in 2-hour PPG from baseline to Week 24 using analysis of covariance model
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 115 | 113
mmol/L | -0.65 [-1.30 to 0.00] | 0.28 [-0.36 to 0.92]
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p = 0.0301, ANCOVA; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.77 to -0.09], Standard Error of Mean 0.426 — Adjusted mean treatment difference from the ANCOVA model (Saxagliptin - Placebo)

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24, Last Observation Carried Forward (LOCF) Measured as [mg/dL]
Description: Adjusted Mean Change in fasting plasma glucose from baseline to Week 24 using analysis of covariance
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 121 | 123
mg/dL | -5.28 [-12.67 to 2.11] | 2.62 [-4.47 to 9.71]
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p = 0.0868, ANCOVA; Mean Difference (Final Values) = -7.90, 95% CI 2-sided [-16.96 to 1.15], Standard Error of Mean 4.595 — Adjusted mean treatment difference from the ANCOVA model (Saxagliptin - Placebo)

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24, Last Observation Carried Forward (LOCF) Measured as [mmol/L]
Description: Adjusted Mean Change in FPG from baseline to Week 24 using analysis of covariance model
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 121 | 123
mmol/L | -0.29 [-0.70 to 0.12] | 0.15 [-0.25 to 0.54]
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p = 0.0868, ANCOVA; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.94 to 0.06], Standard Error of Mean 0.255 — Adjusted mean treatment difference from the ANCOVA model (Saxagliptin - Placebo)

6. Secondary Outcome: Proportion of Participants Achieving a Therapeutic Response: HbA1c Less Than 7% at Week 24, Last Observation Carried Forward (LOCF)
Description: Number of participants achieving a glycaemic response defined as HbA1c less than 7% at Week 24
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - SAXAGLIPTIN | Arm 2 - PLACEBO
Number analyzed (Participants) | 127 | 127
Participants | 39 | 12
Statistical Analysis 1: Comparison: Arm 1 - SAXAGLIPTIN vs Arm 2 - PLACEBO; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 9.006, 95% CI 2-sided [3.852 to 21.05] — Estimated Odds Ratio from the logistic regression model (Saxa/Placebo)

ADVERSE EVENTS:
Arm/Group | SAXAGLIPTIN | PLACEBO
Serious Adverse Events (participants affected / at risk) | 3/129 | 7/128
Other Adverse Events (participants affected / at risk) | 53/129 | 65/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAXAGLIPTIN (N=129) | PLACEBO (N=128)
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAXAGLIPTIN (N=129) | PLACEBO (N=128)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Flatulence (Gastrointestinal disorders) | 4 | 0
Gastritis (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 4
Nasopharyngitis (Infections and infestations) | 8 | 12
Oral Candidiasis (Infections and infestations) | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 6
Urinary Tract Infection (Infections and infestations) | 4 | 8
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 4 | 3
Neuropathy Peripheral (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Hypertension (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submission of any material for publication or presentation, PI shall provide Sponsor with such material for review. If requested in writing by Sponsor, PI shall withhold material from submission for publication or presentation for an additional 90 days from the date of Sponsor's request.